CLINICAL TRIAL: NCT03909178
Title: Arthroscopic Labral Repair Versus Physical Therapy for Tears of the Acetabular Labrum in Patients Age 40 and Older
Brief Title: Arthroscopic Labral Repair Versus Physical Therapy for Tears of the Acetabular Labrum
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Scott D Martin, Principal Investigator, Director, Joint Preservation Service, Director, MGH Sports Medicine Fellowship, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013P001442
Record Dates: First submitted 2018-06-12; First posted 2019-04-09 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Acetabular Labrum Tear; Femoro Acetabular Impingement; Hip Arthroscopy; Physical Therapy; Osteoarthritis, Hip
Keywords: Acetabular Labrum Tear; Femoro Acetabular Impingement; Osteoarthritis; Hip Arthroscopy; Prospective; PROMs; mHHS; HOS; NAHS; LEFS; iHOT-33; RCT, Randomized Control Trial; Physical Therapy, PT; Osteoarthritis, Hip; Tonnis; Outerbridge; Older than 40 years old
MeSH Terms: conditions — Femoracetabular Impingement; Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip Arthroscopy Surgery with Acetabular Labral Repair (Active Comparator): Hip Arthroscopy Surgery with Acetabular Labral Repair
  Interventions: Procedure: Hip Arthroscopy Surgery with Acetabular Labral Repair (SPT group)
- Physical Therapy Focused on the Hip and Hemi-pelvis (Active Comparator): Physical Therapy focusing on the hemipelvis strengthening, including the lower back, lower abdominal core, quadriceps, hamstrings, and gluteal muscles.
  Interventions: Procedure: Physical Therapy Focused on the Hip and Hemi-pelvis (PT group)

INTERVENTIONS:
Procedure: Hip Arthroscopy Surgery with Acetabular Labral Repair (SPT group) — Patients randomized to the SPT group provided consent for arthroscopic acetabular labral repair with femoroacetabular osteoplasty. As previously described in various technique publications from our group, the senior surgeon's (S.D.M.) hip arthroscopy technique includes intra-articular fluid distension for initial portal placement, puncture capsulotomy, autograft capsular augmentation if insufficient or degenerative labral tissue is encountered, intermittent traction, sparing use of electrocautery, and preservation of the chrondrolabral junction. All SPT patients underwent a standardized postoperative physical therapy protocol developed jointly by the senior author (a sports medicine fellowship-trained orthopaedic surgeon) and the physical therapists. Patients were kept weightbearing as tolerated on crutches for 6 weeks to maintain a level pelvis without lurching when walking and were instructed to avoid impact loading exercises for 6 months.
  Arms: Hip Arthroscopy Surgery with Acetabular Labral Repair
Procedure: Physical Therapy Focused on the Hip and Hemi-pelvis (PT group) — PTA patients were assigned a standardized, 24-week course of supervised, core-based PT. This course was designed in concert with physical therapists within our institution to help address symptoms of labral tear in patients older than 40 who had mild to moderate OA. Weeks 1 and 2 focused on normalizing gait, and weeks 3 through 24 focused on optimizing range of motion (ROM) while slowly integrating strength training. Unlike the prerandomization PT protocol, the PTA protocol was predominantly physical therapist-supervised (at least 1 in-person visit per week).
  Arms: Physical Therapy Focused on the Hip and Hemi-pelvis

SUMMARY:
Tears of the acetabular labrum appear to be common with the prevalence of asymptomatic tears in the general population approaching 66% and 70% based on cadaveric dissection and magnetic resonance imaging, respectively. Despite this prevalence, there is no currently accepted justification for performing labral repair in an asymptomatic patient despite the many postulated biomechanical benefits that an intact labrum imparts to the hip joint.

Representing a smaller proportion of all tears, symptomatic tears of the acetabular labrum present a therapeutic challenge. Current treatment modalities range from conservative measures to open surgical intervention. Conservative measures have typically included: activity modification, the use of non-steroidal anti-inflammatory drugs (NSAIDs), physical therapy (PT), core strengthening and improvement of sensory motor control. In the past two decades, technological advances in the form of surgical instrumentation and traction devices have facilitated less invasive arthroscopic techniques to diagnose and treat hip problems and as such is now the preferred treatment modality for many orthopedic surgeons treating patients with hip pathology.

Determining which patients, using age and arthritic burden as predictors, can benefit from labral repair is paramount for several reasons. Showing arthroscopic repair is of little or no benefit to a specific cohort can reduce the number of unnecessary surgeries performed, increase the use of conservative therapy (if validated) and reduce the interval between diagnosis and total hip replacement.

DETAILED DESCRIPTION:
There has been only one prospective study documenting the outcomes of patients treated with physical therapy for intra-articular conditions of the hip. These conditions included mild FAI and mild developmental dysplasia of the hip. Here, physical therapy was given as a first line treatment. Those who did not make satisfactory improvements in pain or wished to have surgery were then scheduled for surgery to repair the defects. Patients saw improvement in validated outcome measures at one year.

Although there have been studies looking at age secondarily in patients with labral tears, there is no prospective evidence to endorse or refute a recommendation of hip arthroscopy for patients of any age being treated for a tear of the acetabular labrum.

Most recently, the authors involved in this study performed a retrospective investigation (unpublished data) to capture patients with clinically and radiographically confirmed acetabular labral pathology electing to undergo conservative management defined as the refusal of surgical intervention. Based on a retrospective review of 894 patients presenting to clinic over a 10-year period, the investigators identified 22 patients with labral pathology that were treated non-operatively. Retrospective case control analysis was performed using outcome questionnaires administered to both surgical and non-surgical cohorts. The investigators found that patients with labral tears managed non-operatively appear to score highly on hip function outcome scores, preliminarily indicating there may be some benefit in using conservative management alone in the treatment of labral pathology.

This is a 12-month prospective randomized control trial (RCT), which will enroll 121 subjects with evidence consistent with a tear of the acetabular labrum. Labral tear will be diagnosed by clinical exam and positive MRI findings. Subjects will receive conservative physical therapy treatment alone or arthroscopic surgical labral repair and physical therapy. The investigators anticipate that pain, range of motion, activity level, and functional performance, as judged by validated outcome measures and serial physical exams, will improve when compared to baseline. The investigators also anticipate that the level of response will be greater in the surgical treatment group than in the physical therapy group at 12 months.

Our Primary Outcome is change in the modified Harris Hip Score at 12 months. Secondary outcomes include changes in other outcomes measures (LEFS, HOS, NAHS, iHOT-33), patient satisfaction, degree of improvement on physical exam, longer-term functional outcomes (i.e., at 2, 5, and 10 years), and the influence of OA severity (Outerbridge scoring) and location on the aforementioned outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 or greater: higher likelihood or undetectable OA on imaging
2. Symptoms consistent with a tear of the acetabular labrum (at least one: catching, clicking, popping, pain with sitting, episodic pain, pain with hip flexion, adduction, and/or internal rotation): asymptomatic labral tears do exist in the general population however there is not definitive evidence to suggest treatment of asymptomatic tears is beneficial.
3. Symptoms not due to some other acute process in or around the hip (including septic arthritis, osteonecrosis, hemarthrosis, iliotibial band syndrome, fractures of the femoral neck or head, fractures of the acetabulum, greater trochanteric pain syndrome, sacroiliac joint pain, piriformis syndrome, low back pain associated with hip pain and not knee nor acute low back injury): certain conditions are not treatable by either arthroscopy or physical therapy. Some of these conditions can be managed with physical therapy but not arthroscopy.
4. Availability of hip radiographs and MRI: needed to assess eligibility
5. Evidence on MRI of a tear of the acetabular labrum: documentation of acetabular labrum tear
6. Willingness to undergo randomization and ability to understand and sign informed consent document: ability to understand study and consent willingly

Exclusion Criteria:

1. Less than 2 mm of joint space on standing plain anterior-posterior radiographs of the hip: indicative of severe osteoarthritic disease and the patient would benefit more from a total hip replacement
2. Developmental dysplasia of the hip: distorted acetabular anatomy and biomechanics
3. Kellgren-Lawrence Grade 4 changes: classified as large osteophytes, marked narrowing of joint space, severe sclerosis, and definite deformity of bone contour; indicative of severe OA
4. Tonnis Grade 3 changes: classified as large cysts in the head or acetabulum, severe narrowing or obliteration of the joint space, severe deformity of the head, and necrosis; indicative of OA
5. Unexpected pathology at the time of arthroscopy: source of pain less likely to due dysfunction of the labrum and more likely due to aberrant extra-articular biology
6. Same site surgery: complex anatomy
7. Back pain greater than hip pain or back pain associated with leg symptoms below the knee: source of pain less likely to be originating from the hip and more likely to be referred from the back/spine
8. Back pain associated with positive neural tension signs e.g. positive slump test, positive SLR (straight leg raise), positive reflex changes or drop foot: source of pain less likely to be originating from the hip and more likely to be referred from the back/spine
9. Knee pain greater than hip pain: source of pain less likely to be originating from the hip and more likely to referred from the knee
10. Bilateral tears of the acetabular labrum: difficult to gauge patient progress after treatment
11. Contraindication to surgery or physical therapy: cannot tolerate either treatment grouping
12. Alternate form of PT for greater than 6 weeks: will negatively augment results. May affect recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-10-21 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2030-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Martin, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH, Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Register B, Pennock AT, Ho CP, Strickland CD, Lawand A, Philippon MJ. Prevalence of abnormal hip findings in asymptomatic participants: a prospective, blinded study. Am J Sports Med. 2012 Dec;40(12):2720-4. doi: 10.1177/0363546512462124. Epub 2012 Oct 25. PMID 23104610
- [Background] Vawklang N, Lertwanich P. Prevalence of acetabular labral tears and sublabral sulci: a cadaveric study. J Med Assoc Thai. 2012 Sep;95 Suppl 9:S104-9. PMID 23326991
- [Background] Alexander JW, Crawford MJ, Vega CE, Thompson MT, Miller AR, Noble PC. The impact of labral tears on the stability of the hip joint. Trans Orthop Res Soc. 2007; 32:71.
- [Background] Crawford MJ, Dy CJ, Alexander JW, Thompson M, Schroder SJ, Vega CE, Patel RV, Miller AR, McCarthy JC, Lowe WR, Noble PC. The 2007 Frank Stinchfield Award. The biomechanics of the hip labrum and the stability of the hip. Clin Orthop Relat Res. 2007 Dec;465:16-22. doi: 10.1097/BLO.0b013e31815b181f. PMID 17906586
- [Background] Song Y, Ito H, Kourtis L, Safran MR, Carter DR, Giori NJ. Articular cartilage friction increases in hip joints after the removal of acetabular labrum. J Biomech. 2012 Feb 2;45(3):524-30. doi: 10.1016/j.jbiomech.2011.11.044. Epub 2011 Dec 15. PMID 22176711
- [Background] Haemer JM, Carter DR, Giori NJ. The low permeability of healthy meniscus and labrum limit articular cartilage consolidation and maintain fluid load support in the knee and hip. J Biomech. 2012 May 11;45(8):1450-6. doi: 10.1016/j.jbiomech.2012.02.015. Epub 2012 Mar 3. PMID 22391467
- [Background] Samora JB, Ng VY, Ellis TJ. Femoroacetabular impingement: a common cause of hip pain in young adults. Clin J Sport Med. 2011 Jan;21(1):51-6. doi: 10.1097/JSM.0b013e318205dfde. PMID 21200171
- [Background] Byrd JW. The role of hip arthroscopy in the athletic hip. Clin Sports Med. 2006 Apr;25(2):255-78, viii. doi: 10.1016/j.csm.2005.12.007. PMID 16638490
- [Background] Enseki KR, Martin RL, Draovitch P, Kelly BT, Philippon MJ, Schenker ML. The hip joint: arthroscopic procedures and postoperative rehabilitation. J Orthop Sports Phys Ther. 2006 Jul;36(7):516-25. doi: 10.2519/jospt.2006.2138. PMID 16881468
- [Background] McCarthy JC, Lee J. Hip arthroscopy: indications and technical pearls. Clin Orthop Relat Res. 2005 Dec;441:180-7. doi: 10.1097/01.blo.0000195057.27653.93. PMID 16331001
- [Background] Groh MM, Herrera J. A comprehensive review of hip labral tears. Curr Rev Musculoskelet Med. 2009 Jun;2(2):105-17. doi: 10.1007/s12178-009-9052-9. Epub 2009 Apr 7. PMID 19468871
- [Background] Khanduja V, Villar RN. Arthroscopic surgery of the hip: current concepts and recent advances. J Bone Joint Surg Br. 2006 Dec;88(12):1557-66. doi: 10.1302/0301-620X.88B12.18584. PMID 17159164
- [Background] Kelly BT, Weiland DE, Schenker ML, Philippon MJ. Arthroscopic labral repair in the hip: surgical technique and review of the literature. Arthroscopy. 2005 Dec;21(12):1496-504. doi: 10.1016/j.arthro.2005.08.013. PMID 16376242
- [Background] Stevens MS, Legay DA, Glazebrook MA, Amirault D. The evidence for hip arthroscopy: grading the current indications. Arthroscopy. 2010 Oct;26(10):1370-83. doi: 10.1016/j.arthro.2010.07.016. PMID 20887936
- [Background] Longo UG, Franceschetti E, Maffulli N, Denaro V. Hip arthroscopy: state of the art. Br Med Bull. 2010;96:131-57. doi: 10.1093/bmb/ldq018. Epub 2010 Jul 6. PMID 20605889
- [Background] Clohisy JC, Keeney JA, Schoenecker PL. Preliminary assessment and treatment guidelines for hip disorders in young adults. Clin Orthop Relat Res. 2005 Dec;441:168-79. doi: 10.1097/01.blo.0000193511.91643.2a. PMID 16331000
- [Background] Safran MR. The acetabular labrum: anatomic and functional characteristics and rationale for surgical intervention. J Am Acad Orthop Surg. 2010 Jun;18(6):338-45. doi: 10.5435/00124635-201006000-00006. PMID 20511439
- [Background] Lewis CL, Sahrmann SA. Acetabular labral tears. Phys Ther. 2006 Jan;86(1):110-21. doi: 10.1093/ptj/86.1.110. No abstract available. PMID 16386066
- [Background] Emara K, Samir W, Motasem el H, Ghafar KA. Conservative treatment for mild femoroacetabular impingement. J Orthop Surg (Hong Kong). 2011 Apr;19(1):41-5. doi: 10.1177/230949901101900109. PMID 21519074
- [Background] Yazbek PM, Ovanessian V, Martin RL, Fukuda TY. Nonsurgical treatment of acetabular labrum tears: a case series. J Orthop Sports Phys Ther. 2011 May;41(5):346-53. doi: 10.2519/jospt.2011.3225. Epub 2011 Feb 18. PMID 21335929
- [Background] Hunt D, Prather H, Harris Hayes M, Clohisy JC. Clinical outcomes analysis of conservative and surgical treatment of patients with clinical indications of prearthritic, intra-articular hip disorders. PM R. 2012 Jul;4(7):479-87. doi: 10.1016/j.pmrj.2012.03.012. Epub 2012 May 16. PMID 22595328
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Background] Kemp JL, Collins NJ, Makdissi M, Schache AG, Machotka Z, Crossley K. Hip arthroscopy for intra-articular pathology: a systematic review of outcomes with and without femoral osteoplasty. Br J Sports Med. 2012 Jul;46(9):632-43. doi: 10.1136/bjsports-2011-090428. Epub 2011 Dec 22. PMID 22194221
- [Background] Larson CM, Giveans MR, Taylor M. Does arthroscopic FAI correction improve function with radiographic arthritis? Clin Orthop Relat Res. 2011 Jun;469(6):1667-76. doi: 10.1007/s11999-010-1741-6. Epub 2010 Dec 22. PMID 21181460
- [Background] Horisberger M, Brunner A, Herzog RF. Arthroscopic treatment of femoral acetabular impingement in patients with preoperative generalized degenerative changes. Arthroscopy. 2010 May;26(5):623-9. doi: 10.1016/j.arthro.2009.09.003. Epub 2010 Feb 11. PMID 20434659
- [Background] Beck M, Kalhor M, Leunig M, Ganz R. Hip morphology influences the pattern of damage to the acetabular cartilage: femoroacetabular impingement as a cause of early osteoarthritis of the hip. J Bone Joint Surg Br. 2005 Jul;87(7):1012-8. doi: 10.1302/0301-620X.87B7.15203. PMID 15972923
- [Background] Beck M, Leunig M, Parvizi J, Boutier V, Wyss D, Ganz R. Anterior femoroacetabular impingement: part II. Midterm results of surgical treatment. Clin Orthop Relat Res. 2004 Jan;(418):67-73. PMID 15043095
- [Background] Jerosch J, Schunck J, Khoja A. Arthroscopic treatment of the hip in early and midstage degenerative joint disease. Knee Surg Sports Traumatol Arthrosc. 2006 Jul;14(7):641-5. doi: 10.1007/s00167-005-0009-2. Epub 2005 Dec 14. PMID 16362355
- [Background] Kim KC, Hwang DS, Lee CH, Kwon ST. Influence of femoroacetabular impingement on results of hip arthroscopy in patients with early osteoarthritis. Clin Orthop Relat Res. 2007 Mar;456:128-32. doi: 10.1097/01.blo.0000246542.49574.2c. PMID 17106273
- [Background] Murphy S, Tannast M, Kim YJ, Buly R, Millis MB. Debridement of the adult hip for femoroacetabular impingement: indications and preliminary clinical results. Clin Orthop Relat Res. 2004 Dec;(429):178-81. doi: 10.1097/01.blo.0000150307.75238.b9. PMID 15577484
- [Background] Margheritini F, Villar RN. The efficacy of arthroscopy in the treatment of hip osteoarthritis. Chir Organi Mov. 1999 Jul-Sep;84(3):257-61. English, Italian. PMID 11569040
- [Background] Philippon MJ, Schroder E Souza BG, Briggs KK. Hip arthroscopy for femoroacetabular impingement in patients aged 50 years or older. Arthroscopy. 2012 Jan;28(1):59-65. doi: 10.1016/j.arthro.2011.07.004. Epub 2011 Oct 7. PMID 21982390
- [Background] McCarthy JC, Jarrett BT, Ojeifo O, Lee JA, Bragdon CR. What factors influence long-term survivorship after hip arthroscopy? Clin Orthop Relat Res. 2011 Feb;469(2):362-71. doi: 10.1007/s11999-010-1559-2. PMID 20872105
- [Background] Hunter DJ. Insights from imaging on the epidemiology and pathophysiology of osteoarthritis. Radiol Clin North Am. 2009 Jul;47(4):539-51. doi: 10.1016/j.rcl.2009.03.004. PMID 19631067
- [Background] von Engelhardt LV, Kraft CN, Pennekamp PH, Schild HH, Schmitz A, von Falkenhausen M. The evaluation of articular cartilage lesions of the knee with a 3-Tesla magnet. Arthroscopy. 2007 May;23(5):496-502. doi: 10.1016/j.arthro.2006.12.027. PMID 17478280
- [Background] Madhusudhan TR, Kumar TM, Bastawrous SS, Sinha A. Clinical examination, MRI and arthroscopy in meniscal and ligamentous knee Injuries - a prospective study. J Orthop Surg Res. 2008 May 19;3:19. doi: 10.1186/1749-799X-3-19. PMID 18489779
- [Background] Fujii M, Nakashima Y, Noguchi Y, Yamamoto T, Mawatari T, Motomura G, Iwamoto Y. Effect of intra-articular lesions on the outcome of periacetabular osteotomy in patients with symptomatic hip dysplasia. J Bone Joint Surg Br. 2011 Nov;93(11):1449-56. doi: 10.1302/0301-620X.93B11.27314. PMID 22058293
- [Background] Streich NA, Gotterbarm T, Barie A, Schmitt H. Prognostic value of chondral defects on the outcome after arthroscopic treatment of acetabular labral tears. Knee Surg Sports Traumatol Arthrosc. 2009 Oct;17(10):1257-63. doi: 10.1007/s00167-009-0833-x. Epub 2009 Jun 30. PMID 19565221
- [Background] Byrd JW, Jones KS. Prospective analysis of hip arthroscopy with 2-year follow-up. Arthroscopy. 2000 Sep;16(6):578-87. doi: 10.1053/jars.2000.7683. PMID 10976117
- [Background] McCormick F, Nwachukwu BU, Alpaugh K, Martin SD. Predictors of hip arthroscopy outcomes for labral tears at minimum 2-year follow-up: the influence of age and arthritis. Arthroscopy. 2012 Oct;28(10):1359-64. doi: 10.1016/j.arthro.2012.04.059. Epub 2012 Aug 17. PMID 22906757
- [Background] Clohisy JC, Carlisle JC, Trousdale R, Kim YJ, Beaule PE, Morgan P, Steger-May K, Schoenecker PL, Millis M. Radiographic evaluation of the hip has limited reliability. Clin Orthop Relat Res. 2009 Mar;467(3):666-75. doi: 10.1007/s11999-008-0626-4. Epub 2008 Dec 2. PMID 19048356
- [Background] Farr J, Cole B, Dhawan A, Kercher J, Sherman S. Clinical cartilage restoration: evolution and overview. Clin Orthop Relat Res. 2011 Oct;469(10):2696-705. doi: 10.1007/s11999-010-1764-z. PMID 21240578
- [Background] Katz JN, Brophy RH, Chaisson CE, de Chaves L, Cole BJ, Dahm DL, Donnell-Fink LA, Guermazi A, Haas AK, Jones MH, Levy BA, Mandl LA, Martin SD, Marx RG, Miniaci A, Matava MJ, Palmisano J, Reinke EK, Richardson BE, Rome BN, Safran-Norton CE, Skoniecki DJ, Solomon DH, Smith MV, Spindler KP, Stuart MJ, Wright J, Wright RW, Losina E. Surgery versus physical therapy for a meniscal tear and osteoarthritis. N Engl J Med. 2013 May 2;368(18):1675-84. doi: 10.1056/NEJMoa1301408. Epub 2013 Mar 18. PMID 23506518
- [Background] Sangha O, Stucki G, Liang MH, Fossel AH, Katz JN. The Self-Administered Comorbidity Questionnaire: a new method to assess comorbidity for clinical and health services research. Arthritis Rheum. 2003 Apr 15;49(2):156-63. doi: 10.1002/art.10993. PMID 12687505
- [Background] Tijssen M, van Cingel R, van Melick N, de Visser E. Patient-Reported Outcome questionnaires for hip arthroscopy: a systematic review of the psychometric evidence. BMC Musculoskelet Disord. 2011 May 27;12:117. doi: 10.1186/1471-2474-12-117. PMID 21619610
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Background] Martin RL, Kelly BT, Philippon MJ. Evidence of validity for the hip outcome score. Arthroscopy. 2006 Dec;22(12):1304-11. doi: 10.1016/j.arthro.2006.07.027. PMID 17157729
- [Background] Martin RL, Philippon MJ. Evidence of reliability and responsiveness for the hip outcome score. Arthroscopy. 2008 Jun;24(6):676-82. doi: 10.1016/j.arthro.2007.12.011. Epub 2008 Mar 12. PMID 18514111
- [Background] Christensen CP, Althausen PL, Mittleman MA, Lee JA, McCarthy JC. The nonarthritic hip score: reliable and validated. Clin Orthop Relat Res. 2003 Jan;(406):75-83. doi: 10.1097/01.blo.0000043047.84315.4b. PMID 12579003
- [Background] Mohtadi NG, Griffin DR, Pedersen ME, Chan D, Safran MR, Parsons N, Sekiya JK, Kelly BT, Werle JR, Leunig M, McCarthy JC, Martin HD, Byrd JW, Philippon MJ, Martin RL, Guanche CA, Clohisy JC, Sampson TG, Kocher MS, Larson CM; Multicenter Arthroscopy of the Hip Outcomes Research Network. The Development and validation of a self-administered quality-of-life outcome measure for young, active patients with symptomatic hip disease: the International Hip Outcome Tool (iHOT-33). Arthroscopy. 2012 May;28(5):595-605; quiz 606-10.e1. doi: 10.1016/j.arthro.2012.03.013. PMID 22542433
- [Background] Griffin DR, Parsons N, Mohtadi NG, Safran MR; Multicenter Arthroscopy of the Hip Outcomes Research Network. A short version of the International Hip Outcome Tool (iHOT-12) for use in routine clinical practice. Arthroscopy. 2012 May;28(5):611-6; quiz 616-8. doi: 10.1016/j.arthro.2012.02.027. PMID 22542434
- [Background] Kopjar B. The SF-36 health survey: a valid measure of changes in health status after injury. Inj Prev. 1996 Jun;2(2):135-9. doi: 10.1136/ip.2.2.135. PMID 9346078
- [Background] Ruta D, Garratt A, Abdalla M, Buckingham K, Russell I. The SF 36 health survey questionnaire. A valid measure of health status.. BMJ. 1993 Aug 14;307(6901):448-9. doi: 10.1136/bmj.307.6901.448-b. No abstract available. PMID 8374477
- [Background] Kellgren JH, Jeffrey MR, Ball J. The Epidemiology of Chronic Rheumatism. Atlas of Standard Radiographs of Arthritis. Oxford, UK: Blackwell Scientific Publications; 1963:vii-11.
- [Background] Tonnis D, Heinecke A, Nienhaus R, Thiele J. [Predetermination of arthrosis, pain and limitation of movement in congenital hip dysplasia (author's transl)]. Z Orthop Ihre Grenzgeb. 1979 Oct;117(5):808-15. German. PMID 549339
- [Background] OUTERBRIDGE RE. The etiology of chondromalacia patellae. J Bone Joint Surg Br. 1961 Nov;43-B:752-7. doi: 10.1302/0301-620X.43B4.752. No abstract available. PMID 14038135
- [Background] Cohen, J. Statistical power analysis for behavioral studies. (2nd ed). New Jersey: Lawrence Erlbaum.
- [Background] Egerton T, Hinman RS, Takla A, Bennell KL, O'Donnell J. Intraoperative cartilage degeneration predicts outcome 12 months after hip arthroscopy. Clin Orthop Relat Res. 2013 Feb;471(2):593-9. doi: 10.1007/s11999-012-2594-y. Epub 2012 Sep 20. PMID 22992870
- [Background] Aprato A, Jayasekera N, Villar RN. Does the modified Harris hip score reflect patient satisfaction after hip arthroscopy? Am J Sports Med. 2012 Nov;40(11):2557-60. doi: 10.1177/0363546512460650. Epub 2012 Sep 28. PMID 23024148
- [Background] Katz JN, Chaisson CE, Cole B, Guermazi A, Hunter DJ, Jones M, Levy BA, Mandl LA, Martin S, Marx RG, Safran-Norton C, Roemer FW, Skoniecki D, Solomon DH, Spindler KP, Wright J, Wright RW, Losina E. The MeTeOR trial (Meniscal Tear in Osteoarthritis Research): rationale and design features. Contemp Clin Trials. 2012 Nov;33(6):1189-96. doi: 10.1016/j.cct.2012.08.010. Epub 2012 Sep 5. PMID 22968127
- [Background] Wilson, S.R. and I. Gordon, Calculating Sample Sizes in the Presence of Confounding Variables. J Royal Statisitical Soc, 1986. 35(2): p. 207-13.
- [Background] Wang R, Lagakos SW, Ware JH, Hunter DJ, Drazen JM. Statistics in medicine--reporting of subgroup analyses in clinical trials. N Engl J Med. 2007 Nov 22;357(21):2189-94. doi: 10.1056/NEJMsr077003. No abstract available. PMID 18032770
- [Derived] Martin SD, Dean MC, Gillinov SM, Cherian NJ, Eberlin CT, Kucharik MP, Abraham PF, Nazal MR, Conaway WK, Quinlan NJ, Alpaugh K, Torabian KA. Hip Arthroscopy Versus Physical Therapy for the Treatment of Symptomatic Acetabular Labral Tears in Patients Older Than 40 Years: 24-Month Results From a Randomized Controlled Trial. Am J Sports Med. 2024 Aug;52(10):2574-2585. doi: 10.1177/03635465241263595. Epub 2024 Aug 5. PMID 39101607
- [Derived] Martin SD, Abraham PF, Varady NH, Nazal MR, Conaway W, Quinlan NJ, Alpaugh K. Hip Arthroscopy Versus Physical Therapy for the Treatment of Symptomatic Acetabular Labral Tears in Patients Older Than 40 Years: A Randomized Controlled Trial. Am J Sports Med. 2021 Apr;49(5):1199-1208. doi: 10.1177/0363546521990789. Epub 2021 Mar 3. PMID 33656950

RESULTS

PARTICIPANT FLOW:
Groups:
- Hip Arthroscopy Surgery With Acetabular Labral Repair: Hip Arthroscopy Surgery with Acetabular Labral Repair
  Hip Arthroscopy Surgery with Acetabular Labral Repair: The research coordinator will, perform a baseline assessment, and randomize the patients into the study at this visit.
  Randomization will be assigned utilizing an electronic randomization program. Patients are prospectively identified and randomized into one of two study arms: arthroscopic surgery (AS) or physical therapy (PT). A third study arm, dependent upon improvement with PT, was created as patients crossed over (CO) from PT to AS after a lack of improvement after a minimum of 8 weeks of PT. AS consisted of labral repair.
  Any subject randomized to surgery will be seen by Dr. Martin to be consented separately for the arthroscopic procedure, which is standard of care. Those receiving surgical management will be scheduled for the post-operative physical therapy protocol within 2 weeks of their operative date, once a surgical date has been scheduled.
- Physical Therapy Focused on the Hip and Hemi-pelvis: Physical Therapy focusing on the hemipelvis strengthening, including the lower back, lower abdominal core, quadriceps, hamstrings, and gluteal muscles.
  Physical Therapy Focused on the Hip and Hemi-pelvis: The research coordinator will, perform a baseline assessment, and randomize the patients into the study at this visit.
  Randomization will be assigned utilizing an electronic randomization program. Patients are prospectively identified and randomized into one of two study arms: arthroscopic surgery (AS) or physical therapy (PT). A third study arm, dependent upon improvement with PT, was created as patients crossed over (CO) from PT to AS after a lack of improvement after a minimum of 8 weeks of PT. AS consisted of labral repair or debridement, if repair was not possible, and PT consisted of a uniform, comprehensive PT protocol guided by selected physical therapists.
  Those randomized to the physical therapy side will be referred to PT. Those receiving conservative management will be scheduled for physical therapy.
Period: Overall Study
Arm/Group | Hip Arthroscopy Surgery With Acetabular Labral Repair | Physical Therapy Focused on the Hip and Hemi-pelvis
Started | 57 | 53
Completed | 54 | 49
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- SPT Group: Surgery and Physical Therapy: Patients randomized to the SPT group provided consent for arthroscopic acetabular labral repair with femoroacetabular osteoplasty. As previously described in various technique publications from our group, the senior surgeon's (S.D.M.) hip arthroscopy technique includes intra-articular fluid distension for initial portal placement,2 puncture capsulotomy,9 autograft capsular augmentation if insufficient or degenerative labral tissue is encountered,28,30 intermittent traction,37 sparing use of electrocautery,24 and preservation of the chrondrolabral junction.39 All SPT patients underwent a standardized postoperative physical therapy protocol developed jointly by the senior author (a sports medicine fellowship-trained orthopaedic surgeon) and the physical therapists. Patients were kept weightbearing as tolerated on crutches for 6 weeks to maintain a level pelvis without lurching when walking and were instructed to avoid impact loading exercises for 6 months. Appendix A (available in the online version of this article) provides the complete postoperative physical therapy protocol.
- PTA Group: Physical Therapy Alone: PTA patients were assigned a standardized, 24-week course of supervised, core-based PT. This course was designed in concert with physical therapists within our institution to help address symptoms of labral tear in patients older than 40 who had mild to moderate OA. Weeks
  1 and 2 focused on normalizing gait, and weeks 3 through 24 focused on optimizing range of motion (ROM) while slowly integrating strength training. Unlike the prerandomization PT protocol, the PTA protocol was predominantly physical therapist-supervised (at least 1 in-person visit per week. Appendix B (available online) provides the complete 24- week PT protocol assigned to PTA patients.
- Total: Total of all reporting groups
Arm/Group | SPT Group: Surgery and Physical Therapy | PTA Group: Physical Therapy Alone | Total
Number analyzed (Participants) | 57 | 53 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 56 | 53 | 109
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 49.6 [40 to 67] | 49.1 [40 to 67] | 49.4 [40 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 30 | 62
  Male | 25 | 23 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 53 | 47 | 100
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 46 | 44 | 90
Radiographic Osteoarthritis [Mean (Inter-Quartile Range); unit: units on a scale] — Tonnis grading is used to evaluate the extent of hip osteoarthritis seen on a plain anterior-posterior radiograph. Radiographs were graded by fellowship trained musculoskeletal radiologists. The scale is from 0-3 and is shown below.
  0: no signs of osteoarthritis
  1. minor joint space narrowing, subchondral sclerosis of the femoral head and/or acetabulum, small osteophytes
  2. moderate joint space narrowing, small subchondral cysts, moderate loss of sphericity of the femoral head
  3. severe joint space narrowing or obliteration, large subchondral cysts, severe deformity of the femoral head
  units on a scale | 1.22 [1.09 to 1.34] | 1.27 [1.12 to 1.42] | 1.24 [1.14 to 1.34]
Body Mass Index [Mean (Inter-Quartile Range); unit: kg/m^2] | 27.1 [25.8 to 28.4] | 26.8 [25.6 to 28.0] | 26.9 [26.1 to 27.8]
modified Harris Hip Score [Mean (Inter-Quartile Range); unit: units on a scale] — The modified Harris Hip Scale (mHHS) was developed for the assessment of the results of hip surgery, and is intended to evaluate various hip disabilities and methods of treatment in an adult population. It features a series of questions that are subjectively completed by the patient, which provides a value output (higher score = better result). The interpretation of outcome using the modified Harris hip score was as follows: <70 (poor result), 70-79 (fair result), 80-89 (good result) and >90 (excellent result).
  units on a scale | 65.3 [61.4 to 69.1] | 63 [59 to 67] | 64.2 [61.4 to 66.9]
VAS Pain Score [Mean (Inter-Quartile Range); unit: units on a scale] — The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain." Higher values = higher pain and worse outcome. Absolute values of pain on a 0-10 scale naturally grouped into three categories: 1-4 (mild pain), 5 or 6 (moderate pain) and 7-10 (severe pain).
  units on a scale | 6.2 [5.5 to 6.9] | 6.0 [5.2 to 6.7] | 6.1 [5.6 to 6.6]
International Hip Outcome Tool - 33 [Mean (Inter-Quartile Range); unit: units on a scale] — The International Hip Outcome Tool (iHOT) was developed by Mohtadi et al as a means of assessing a patient's ability to return to an active lifestyle through obtaining subjective measures of symptoms, as well as determining emotional and social health status. The iHOT is comprised of 33 questions relating to: Symptoms and Functional Limitations, Sports and Recreational Activities, Job-Related Concerns, Social, Emotional, and Lifestyle Concerns. Higher scores = better function and less limitations.
  units on a scale | 38.9 [33.9 to 43.9] | 37 [31.6 to 42.4] | 38.0 [34.4 to 41.6]

OUTCOME MEASURES:

1. Primary Outcome: Change in mHHS Surveys From Preoperative to Various Postoperative Timepoints
Description: Full Name of Outcome: modified Harris Hip Score (mHHS)
  Purpose: Validated Hip Patient Reported Outcome Measurements (PROMs) to assess the patient's functional outcomes post-surgery.
  Scale of mHHS:
  Min: 0 Max: 100
  Higher score indicates better hip functionally.
  No subscores or subscales.
  The mean changes in scores required to achieve a minimically clinically important difference is 6.9.
Time Frame: Baseline (pre-operative), 3 months, 6 months, 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- PTA Group: Physical Therapy Alone Group: PTA patients were assigned a standardized, 24-week course of supervised, core-based PT. This course was designed in concert with physical therapists within our institution to help address symptoms of labral tear in patients older than 40 who had mild to moderate OA. Weeks
  1 and 2 focused on normalizing gait, and weeks 3 through 24 focused on optimizing range of motion (ROM) while slowly integrating strength training. Unlike the prerandomization PT protocol, the PTA protocol was predominantly physical therapist-supervised (at least 1 in-person visit per week. Appendix B (available online) provides the complete 24- week PT protocol assigned to PTA patients.
Arm/Group | SPT Group: Surgery and Physical Therapy | PTA Group: Physical Therapy Alone Group
Number analyzed (Participants) | 42 | 39
units on a scale
  mHHS improvement at 3 months | 9.26 [8.13 to 10.5] | 4.42 [3.66 to 5.18]
  mHHS improvement at 6 months | 12.63 [11.56 to 13.8] | 6.98 [6.24 to 7.72]
  mHHS improvement 12 months | 17.32 [16.12 to 18.62] | 12.63 [12.27 to 12.99]

2. Secondary Outcome: Change HOS Surveys From Preoperative to Various Postoperative Timepoints
Description: Full Name of Outcome: HOS--Hip Outcome Score.
  Purpose: Validated Hip Patient Reported Outcome Measurements (PROMs) to assess the patient's functional outcomes post-surgery.
  Scale of HOS:
  Min: 0 Max: 100
  No standardized scoring categories (i.e. excellent, good, fair, poor).
  Higher score indicates better hip functionally.
  The mean change in HOS score required to achieve a minimally clinically important difference is 8.8.
Time Frame: Baseline (pre-operative), 3 months, 6 months, 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Hip Arthroscopy Surgery With Acetabular Labral Repair | Physical Therapy Focused on the Hip and Hemi-pelvis
Number analyzed (Participants) | 46 | 44
units on a scale
  HOS improvement at 3 Months | 13.36 [8.21 to 18.51] | 8.44 [3.58 to 13.30]
  HOS improvement at 6 Months | 17.04 [11.95 to 22.13] | 8.36 [3.57 to 13.15]
  HOS improvement at 12 Months | 20.22 [15.00 to 25.43] | 15.07 [10.65 to 19.49]

3. Secondary Outcome: Change NAHS Surveys From Preoperative to Various Postoperative Timepoints
Description: Full Name of Outcome: Non-Arthritic Hip Score (NAHS)
  Purpose: Validated Hip Patient Reported Outcome Measurements (PROMs) to assess the patient's functional outcomes post-surgery:
  Scale of NAHS:
  Min: 0 Max: 100
  No standardized scoring categories (i.e. excellent, good, fair, poor).
  Higher score indicates better hip functionally.
  No subscores or subscales.
  No specific score to indicate a minimally clinically important difference.
Time Frame: Baseline (pre-operative), 3 months, 6 months, 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SPT Group: Surgery and Physical Therapy | PTA Group: Physical Therapy Alone Group
Number analyzed (Participants) | 46 | 44
units on a scale
  3 Months improvement NAHS score | 12.91 [7.58 to 17.30] | 5.26 [0.57 to 9.95]
  6 Months improvement NAHS score | 19.40 [14.45 to 24.36] | 8.68 [4.06 to 13.29]
  12 Months improvement NAHS score | 21.88 [16.79 to 26.96] | 14.94 [10.56 to 19.32]

4. Secondary Outcome: Change iHOT--33 Surveys From Preoperative to Various Postoperative Timepoints
Description: Full Name of Outcome: International Hip Outcome Tool--33 Questions
  Purpose: Validated Hip Patient Reported Outcome Measurements (PROMs) to assess the patient's functional outcomes post-surgery.
  Scale of iHOT-33:
  Min: 0 Max: 100
  No standardized scoring categories (i.e. excellent, good, fair, poor).
  Higher score indicates better hip functionally.
  No subscores or subscales
  The mean changes in iHOT-33 scores required to achieve minimally clinically important difference is 15.1.
Time Frame: Baseline (pre-operative), 3 months, 6 months, 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SPT Group: Surgery and Physical Therapy | PTA Group: Physical Therapy Alone Group
Number analyzed (Participants) | 46 | 44
units on a scale
  3 Months iHOT improvement | 18.37 [10.59 to 24.14] | 4.53 [-1.69 to 10.76]
  6 Months iHOT improvement | 25.28 [18.59 to 31.96] | 13.23 [7.09 to 19.37]
  12 Months iHOT improvement | 33.55 [26.85 to 40.24] | 20.53 [14.76 to 26.30]

5. Secondary Outcome: Change LEFS Surveys From Preoperative to Various Postoperative Timepoints
Description: Full Name of Outcome: Lower Extremity Functional Scale (LEFS)
  Purpose: Validated Hip Patient Reported Outcome Measurements (PROMs) to assess the patient's functional outcomes post-surgery.
  Scale of LEFS:
  Min: 0 Max: 100
  No standardized scoring categories (i.e. excellent, good, fair, poor).
  Higher score indicates better hip functionally.
  There is no designated improvement that is deemed to be a minimally clinically important difference
Time Frame: Baseline (pre-operative), 3 months, 6 months, 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SPT Group: Surgery and Physical Therapy | PTA Group: Physical Therapy Alone Group
Number analyzed (Participants) | 46 | 44
units on a scale
  3 Months improvements LEFS | 6.74 [2.13 to 11.36] | 5.11 [0.81 to 9.42]
  6 Months improvements LEFS | 15.61 [11.05 to 20.17] | 6.77 [2.53 to 11.01]
  12 Months improvements LEFS | 18.46 [13.78 to 23.14] | 12.18 [8.18 to 16.19]

6. Secondary Outcome: Degree of Improvement on Hip VAS Pain Score
Description: At routine follow-up visits patients will be asked to rate hip pain using the VAS (Visual Analog Scale) Score
  Min: 0--no pain Max: 10--worst pain experienced in their life
  Increments of 1.
  Categories:
  1--3: mild pain 4--6: moderate pain 7--10: severe pain
  There is no reduction in VAS score that is considered a minimally clinically important difference.
Time Frame: Baseline (pre-operative), 3 months, 6 months, 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SPT Group: Surgery and Physical Therapy | PTA Group: Physical Therapy Alone Group
Number analyzed (Participants) | 46 | 44
units on a scale
  3 Months VAS change | 3.02 [2.21 to 3.83] | 1.05 [0.24 to 1.86]
  6 Months VAS change | 3.67 [2.96 to 4.39] | 0.79 [-0.13 to 1.71]
  12 Months VAS change | 3.51 [2.92 to 4.09] | 2.21 [0.78 to 3.63]

ADVERSE EVENTS:
Time Frame: 2 years. Each patient is followed clinically by the provider for 2 years from the time of enrollment into the study.
Description: The definitions do not differ.
Groups:
- SPT Group: Surgery and Physical Therapy: Patients randomized to the SPT group provided consent for arthroscopic acetabular labral repair with femoroacetabular osteoplasty. As previously described in various technique publications from our group, the senior surgeon's (S.D.M.) hip arthroscopy technique includes intra-articular fluid distension for initial portal placement, puncture capsulotomy, autograft capsular augmentation if insufficient or degenerative labral tissue is encountered, intermittent traction, sparing use of electrocautery, and preservation of the chrondrolabral junction. All SPT patients underwent a standardized postoperative physical therapy protocol developed jointly by the senior author (a sports medicine fellowship-trained orthopaedic surgeon) and the physical therapists. Patients were kept weightbearing as tolerated on crutches for 6 weeks to maintain a level pelvis without lurching when walking and were instructed to avoid impact loading exercises for 6 months.
Arm/Group | SPT Group: Surgery and Physical Therapy | PTA Group: Physical Therapy Alone.
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/44
Other Adverse Events (participants affected / at risk) | 0/46 | 0/44

LIMITATIONS AND CAVEATS:
Crossover rates in this study were high. For ethical reasons, all randomized patients had to meet surgical eligibility, potentially increasing crossover rates because participants randomized to PTA were aware that they met surgical eligibility. Second, some patients may have had bias for either SPT or PTA. However, to minimize this bias, we imposed strict inclusion criteria to ensure that patients did not prefer one treatment arm and were fully committed to completing their assigned treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT03909178/Prot_SAP_ICF_000.pdf